CLINICAL TRIAL: NCT01738464
Title: Microbiomes of Pelvic Pain
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: STU00055668; 1R01DK103769-01A1 (NIH)
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Interstitial Cystitis; Chronic Prostatitis; Chronic Pelvic Pain Syndrome; Lower Urinary Tract Symptoms; Overactive Bladder; Major Depression
Keywords: Pelvic Pain; Interstitial Cystitis; Microbiome; Prostatitis; Chronic; Depression
MeSH Terms: conditions — Cystitis, Interstitial; Lower Urinary Tract Symptoms; Urinary Bladder, Overactive; Depressive Disorder, Major; Pelvic Pain; Prostatitis; Bronchiolitis Obliterans Syndrome; Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool specimen, Blood/Serum specimen, Urine specimen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pelvic Pain: Interstitial Cystitis or Chronic Prostatitis/Chronic Pelvic Pain Syndrome, Lower Urinary Tract Symptoms, and Overactive Bladder patients will be compared to Healthy and Depressed patients.
- Controls: Healthy patients will be used as controls to compare to patients diagnosed with Interstitial Cystitis, Chronic Prostatitis, Chronic Pelvic Pain Syndrome, Lower Urinary Tract Symptoms, Overactive Bladder, and Depressed patients.
- Major Depression: Major Depression patients will be compared to Controls and Pelvic Pain cohorts.

SUMMARY:
This research study seeks to provide more insight as to how the microbiome affects or is affected by conditions causing chronic pelvic pain such as Interstitial Cystitis (IC), Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS), Lower Urinary Tract Symptoms (LUTS), or Overactive bladder (OAB). Depression and many chronic pain disorders are often related and are poorly understood, and treatment is often not helpful. The goal of this study is to explain pelvic pain characteristics and causes by studying microbiomes of healthy people compared to people suffering from IC, CP/CPPS, LUTS, OAB, and Major depression.

DETAILED DESCRIPTION:
Interstitial cystitis/painful bladder syndrome (IC) or Chronic Prostatitis/Chronic Pelvic Pain Syndrome (CP/CPPS) is characterized by chronic pelvic pain and voiding dysfunction. IC or CP/CPPS remains an enigma within urology, with no known etiology or widely effective therapies. However, some IC, CP/CPPS, and depressed patients suffer bowel co-morbidities, and it is well established that the GI tract can influence bladder function, mood and sensation via pelvic organ crosstalk. Like other body sites, the gut harbors a rich microflora. Studies characterizing microbial diversity and relative abundance at a particular body site, the "microbiome," reveal that microbiomes play critical roles in normal cellular and organ function, and thus this importance is emphasized with the Human Microbiome Project (HMP), an NIH Common Fund initiative. CPPS patients suffer chronic pelvic pain and dramatically lower quality of life, yet diagnostic markers and effective therapies remain elusive for these costly syndromes. IC is a debilitating condition of pelvic pain and voiding dysfunction afflicting up to 8 million U.S. women where depression is a common co-morbidity, distinct from over-active bladder (OAB) patients lacking pain. IC etiology remains unknown, but urothelial lesions and lamina propria mast cells are associated with patient symptoms. Similarly, CP/CPPS afflicts 1 in 22 men in the U.S. with pain and voiding and sexual symptoms, again distinct from patients having only irritative voiding from lower urinary tract symptoms (LUTS). And although leukocytes are observed in prostatic fluid of some patients, the etiology of CP/CPPS also remains unknown. Hypothalamic-pituitary-adrenal axis (HPA) dysfunction has been implicated in female and male patients and cats with feline IC, and thus may be common among CPPS, but a mechanism that integrates pelvic pain, voiding dysfunction, HPA activity, and depression is lacking.

Microbiomes are also dynamic and subject to skewing, and these changes are increasingly associated with diseases including Crohn's disease, ulcerative colitis, obesity, and possibly depression. Antibiotic therapies alter microbiomes, often causing temporary dysfunction and sometimes resulting in diseases such as colitis. Since IC or CP/CPPS patients often have a history of urinary tract infection (UTI), they typically receive multiple courses of antibiotics. This therapeutic history of IC or CP/CPPS patients may have adverse consequences for two reasons. First, potential skewing of the gut microbiome may alter normal sensory and functional homeostatic mechanisms, contributing to pain and voiding dysfunction. Second, an altered gut microbiome may foster uropathogen reservoir expansion, and our preliminary data demonstrate urinary E. coli isolates can induce chronic pelvic pain persisting long after microbial clearance. Together these lines of reasoning raise the provocative possibility that microbiomes contribute to IC, CP/CPPS, and depression directly by supplying uropathogens or indirectly through organ crosstalk dysfunction. Therefore, is an altered gastrointestinal tract microbiome associated with IC, CP/CPPS, and/or depression? Our team marries core NIH and NIDDK missions, digestive diseases and kidney/urologic, to address this novel question with synergistic expertise in clinical diagnosis of IC, CP/CPPS, and depression, quantifying GI tract microbiomes, and neural mechanisms of microbe-induced pelvic pain. Stool samples will be analyzed by 16S rDNA sequence and in silico metagenome analyses to identify taxa, abundance, and function. Computational tools will be used to identify taxa amenable to rapid evaluation of stool. Stool, serum, and urine will be evaluated for small molecules specific to CPPS, and these putative mediators will be tested in mice for effects on pelvic pain and urinary function.

ELIGIBILITY:
Inclusion Criteria:

* Any sex
* Between the ages of 18 and 60
* Any ethnicity
* Have provided informed consent
* Physician diagnosis of interstitial cystitis/bladder pain syndrome (IC/BPS), interstitial cystitis/painful bladder syndrome (IC/PBS), chronic prostatitis/chronic pelvic pain syndrome (CP/CPPS), Lower Urinary Tract Symptoms, Overactive Bladder, or Major Depression.
* Report symptoms of discomfort or pain in the pelvic or abdominal region of moderate severity for at least a three (3) month period within the last six (6) months, who have been currently diagnosed with major depression
* Are healthy, age matched, controls.

Exclusion Criteria:

For IC/CPPS/LUTS/OAB

* Evidence of facultative Gram negative or enterococcus with a value of ≥ 100,000 colony forming units (CFU)/milliliter in mid-stream urine (VB2)
* Secondary chronic pain condition which would prevent a clear interpretation of the study results
* A history of tuberculous cystitis, bladder cancer, carcinoma in situ, or urethral cancer; history of alcohol abuse, inflammatory bowel disease, pelvic radiation or systemic chemotherapy, intravesical chemotherapy, intravesical Bacillus Calmette-Guerin (BCG), active urethral stricture, ureteral calculi, urethral diverticulum, or neurological disease or disorder affecting the bladder or gut
* Unlikely to be compliant due to unmanaged medical or psychological conditions, including neurological, psychological or speech/language problems that will interfere or prevent with their understanding of consent
* Ability to comply with the protocol or ability to complete the study
* Pregnant or Syndromes of Chronic Pelvic Pain (SCPP) symptoms are present only during menses
* And if there was antibiotic use in the last 6 months

For Depressed Patients:

* Participant is in remission or has recovered from major depression, has substance abuse in the past 6 months, has been diagnosed with any bipolar or psychotic disorder, has been diagnosed with any severe cognitive impairment or dementia, history of cancer (with the exception of skin cancer), has current major psychiatric disorder or other psychiatric or medical comorbidities that would interfere with study participation (e.g. dementia, psychosis, upcoming major surgery, lupus, active heart failure, diabetes, etc., currently has a UTI and/or has had a positive urine culture in the past 6 weeks, and if there was antibiotic use in the last 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Primary care clinic patients Community sample
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2012-06; Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-08 (Actual)

PRIMARY OUTCOMES:
Genotype Anaerobic Bacterial populations between Control patients and patients diagnosed with Interstitial Cystitis or Chronic Prostatitis/Chronic Pelvic Pain Syndrome, Lower Urinary Tract Symptoms, Overactive Bladder, and Major Depression | 1 day
  Anaerobic bacteria will be collected from a fecal specimen from both Control patients and patients diagnosed with Interstitial Cystitis or Chronic Prostatitis/Chronic Pelvic Pain Syndrome, Lower Urinary Tract Symptoms, Overactive Bladder, and/or Major Depression. Genotyping will be done to differentiate bacterial populations between the Control patients and patients with Interstitial Cystitis or Chronic Prostatitis/Chronic Pelvic Pain Syndrome, Lower Urinary Tract Symptoms, Overactive Bladder, and/or Major Depression.
Separate serum from blood specimen given by Control patients and patients diagnosed with Interstitial Cystitis or Chronic Prostatitis/Chronic Pelvic Pain Syndrome, Lower Urinary Tract Symptoms, Overactive Bladder, and Major Depression | 3 days
  If you are a local patient: Blood will be collected and serum will be separated and analyzed for HPA markers associated with the anaerobic organisms found in the microbiome.
Collect urine specimen from Control patients and patients diagnosed with Interstitial Cystitis or Chronic Prostatitis/Chronic Pelvic Pain Syndrome, Lower Urinary Tract Symptoms, Overactive Bladder, and Major Depression | 3 days
  If you are a local patient: Urine will be analyzed for the presence of bacteria, and HPA markers associated with the organisms found in the microbiome.

CONTACTS AND LOCATIONS:
Overall Officials: David J Klumpp, PhD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States